CLINICAL TRIAL: NCT06701643
Title: Can Neutrophil-to-Lymphocyte Ratio, Platelet Volume and Platelet Distribution Width Be Used as Indicators of Delirium?
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E1-23-3197
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Delirium - Postoperative
Keywords: postoperative delirium; children; general anesthesia; neutrophil-to-lymphocyte ratio
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing adenoidectomy, tonsillectomy and/or ventilation tube application: Patients undergoing adenoidectomy, tonsillectomy and/or ventilation tube application either premedicated or not, with ASA I-III risk group, followed up for 30 minutes postoperatively.

SUMMARY:
Postoperative delirium is a frequent complication in children undergoing general anesthesia. It has been suggested that inflammation and oxidative stress contribute to the pathophysiology of delirium. The aim of this prospective observational study was to investigate the relationship between inflammatory markers, and delirium. The main questions it aimed to answer were:

* Is there a realtionship between delirium and neutrophil-to-lymphocyte ratio?
* Is there a realtionship between delirium and platelet volume?
* Is there a realtionship between delirium and platelet distribution width?
* What is the incidence of postoperative delirium in the study group?

DETAILED DESCRIPTION:
Postoperative delirium is a frequent complication in children undergoing general anesthesia. It has been suggested that inflammation and oxidative stress contribute to the pathophysiology of delirium. The aim of our study was to investigate the relationship between inflammatory markers, and delirium.

This single-center, prospective, and observational study included 221 children aged 3 to 9 years in the ASA 1-3 risk group who underwent adenoidectomy, tonsillectomy, and/or ventilation tube placement. Consent was obtained from the parents, and patients were either premedicated with oral midazolam in the preoperative period or taken to surgery without premedication, depending on the anesthesiologist's preference. After induction with sevoflurane, intravenous access was established, and fentanyl (1 µg.kg-1) and rocuronium (0.6 mg.kg-1) were administered. Following intubation, maintenance was achieved with sevoflurane, 50% oxygen, 50% air, and a remifentanil infusion at 0.1-0.15 µg.kg-1.min-1. Additionally, all children received intravenous paracetamol (15 mg.kg-1), methylprednisolone (1 mg.kg-1), and ondansetron (0.1 mg.kg-1). At the end of the operation, the muscle relaxant effect was reversed with sugammadex at 2 mg.kg-1. Following extubation, patients were transferred to the post-anesthesia recovery unit and monitored for 30 minutes in the presence of their parents. In the postoperative period, patients' pain was assessed using the Face, Legs, Activity, Cry, and Consolability (FLACC) Scale, and the presence of delirium was evaluated with the Pediatric Anesthesia Emergence Delirium (PAED) Scale.

The FLACC Scale is used to assess the intensity of postoperative pain in young children, infants, or those unable to communicate. Each parameter is assessed on a scale from 0 to 2, with the total score interpreted as follows: 0 = relaxed and comfortable, 1-3 = mild discomfort, 4-6 = moderate pain, and 7-10 = severe discomfort/pain. A score greater than 3 indicates a need for analgesics In our study, ibuprofen was administered to patients experiencing pain within the first 30 minutes of the postoperative period.

The Pediatric Anesthesia Emergence Delirium (PAED) Scale is the only validated tool for measuring delirium and agitation in the postoperative period. The PAED score is used to assess delirium after the patient awakens and prior to the administration of medication, in order to differentiate pain from delirium. Accordingly, the PAED score is determined by evaluating each category-eye contact, purposeful movements, awareness of surroundings, restlessness, and inconsolability-on a scale from 0 to 4. A total score equal to or greater than 10 indicates the presence of delirium. In our study, all patients were assessed using the PAED scoring system in the postoperative period, and those with a score of 10 or higher were considered to have delirium.

Complete blood count values that are routinely measured in the preoperative period were recorded for all patients.

Statistical analysis Data analysis was performed using the R Studio package program (RStudio Team (2020), Integrated Development for R. RStudio, PBC, Boston, MA, http://www.rstudio.com/ ). In our descriptive analyses, quantitative data were expressed as mean and standard deviation, while qualitative categorical variables were presented as case numbers and percentages (%). In the analysis of NLR levels in patients classified as having delirium, tests for normal distribution and homogeneity of variance were conducted to ensure the assumptions for the Student's t-test were met. Shapiro-Wilk normality tests were performed for the "Yes" and "No" groups. The Student's t-test was used to compare the mean NLR levels between the two groups. The association between the need for analgesics and the presence of delirium in children was evaluated using the Pearson chi-square test with Yates continuity correction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III risk group
* Planned to have adenoidectomy, tonsillectomy, and/or ventilation tube placement.

Exclusion Criteria:

* Children under 3 years old
* Children over 9 years old

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This single-center study, took place in Ankara Bilkent City Hospital's operating rooms and postoperative care unit. Children undergoing adenoidectomy, tonsillectomy, and/or ventilation tube placement were followed up.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Neutrophil-to-lymphocyte ratio in the study group including patients with and without delirium | Preoperatively, at the preoperative assessment
  Preoperative Neutrophil-to-lymphocyte ratio recorded from routine preoperative blood tests.
Platelet volume in the study group including patients with and without delirium | Preoperatively, at the preoperative assessment
  Preoperative Platelet volume recorded from routine preoperative blood tests.
Platelet Distribution Width in the study group including patients with and without delirium | Preoperatively, at the preoperative assessment
  Preoperative Platelet Distribution Width recorded from routine preoperative blood tests.
Incidence of postoperative delirium | 30 minutes postoperatively
  Patients are followed up for 30 minutes postoperatively and delirium is detected via The Pediatric Anesthesia Emergence Delirium (PAED) Score. PAED score is determined by evaluating each category-eye contact, purposeful movements, awareness of surroundings, restlessness, and inconsolability-on a scale from 0 to 4. A total score equal to or greater than 10 indicates the presence of delirium (. In our study, all patients were assessed using the PAED scoring system in the postoperative period, and those with a score of 10 or higher were considered to have delirium.

SECONDARY OUTCOMES:
Incidence of postoperative pain | 30 minutes postoperatively
  Patients are followed up for 30 minutes postoperatively and patients' pain was assessed using the Face, Legs, Activity, Cry, and Consolability (FLACC) Scale. The FLACC Scale is used to assess the intensity of postoperative pain in young children, infants, or those unable to communicate. Each parameter is assessed on a scale from 0 to 2, with the total score interpreted as follows: 0 = relaxed and comfortable, 1-3 = mild discomfort, 4-6 = moderate pain, and 7-10 = severe discomfort/pain. A score greater than 3 indicates a need for analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Erkilic, Associate Professor, Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology
Locations (1):
- Ankara Bilkent City Hospital, Department of Anesthesiology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after publication of the study. Study protocol, statistical analysis, study report will be shared if required by a researcher.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning right after publication and ending 2 years after the publication of results
Access Criteria: Data required for researches will be shared

REFERENCES:
- [Result] Ida M, Takeshita Y, Kawaguchi M. Preoperative serum biomarkers in the prediction of postoperative delirium following abdominal surgery. Geriatr Gerontol Int. 2020 Dec;20(12):1208-1212. doi: 10.1111/ggi.14066. Epub 2020 Oct 21. PMID 33084189
- [Result] Vlajkovic GP, Sindjelic RP. Emergence delirium in children: many questions, few answers. Anesth Analg. 2007 Jan;104(1):84-91. doi: 10.1213/01.ane.0000250914.91881.a8. PMID 17179249
- [Result] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Result] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952
- [Result] Feng B, Guo Y, Tang S, Zhang T, Gao Y, Ni X. Association of preoperative neutrophil-lymphocyte ratios with the emergence delirium in pediatric patients after tonsillectomy and adenoidectomy: an observational prospective study. J Anesth. 2024 Apr;38(2):206-214. doi: 10.1007/s00540-023-03303-3. Epub 2024 Jan 24. PMID 38267728
- [Result] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810